CLINICAL TRIAL: NCT03236831
Title: AKI Prevention and Early Intervention in Patients Undergoing VAD Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Qi Qian, M.D., Professor of Medicine and Physiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-001893
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Kidney Injury
Keywords: Ventricular Assist Device

STUDY DESIGN:
Intervention Model Description: Open label single group interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects Undergoing Prospective VAD (Other): Patients undergoing VAD placement. The investigators will provide clinical recommendations to the subject's primary care provider.
  Interventions: Other: Clinical Recommendations

INTERVENTIONS:
Other: Clinical Recommendations — The investigators will provide clinical recommendations to the subject's primary care provider. These will be in regards to the following:
  1. Avoidance of potentially nephrotoxic medications.
  2. Optimizing volume status (avoidance of volume overload or depletion)
  3. Optimizing electrolytes and acid-base status
  4. Minimizing IV contrast exposure when appropriate
  5. Treating severe anemia
  6. Optimization of hemodynamics (Mean arterial BP>65mmHg)

SUMMARY:
The investigators are doing this research to find out if more careful assessment and elimination of potential risk factors of acute kidney injury (AKI) during the subject's perioperative period will reduce their chance of kidney damage and kidney damage related problems.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether preventive measures for patients undergoing ventricular assist device (VAD) placement will reduce AKI occurrence, progression and associated complications.

Participants will be in the study for a total of 6 days (1 day prior to the surgery and 5 days after the surgery). The investigators will review the participant's medical record up to one year after surgery.

The study investigators will access the participant's electronic medical record 24 hours prior to the planned VAD implantation and review the participant's medication regimen and provide recommendations to the participant's primary care physician in an effort to minimize potential risks for AKI. There will be no intervention during the operation.

The clinical recommendations will cover the following:

1. Avoidance of potentially nephrotoxic agents.
2. Optimizing volume status (avoidance of volume overload or depletion)
3. Optimizing electrolytes and acid-base status
4. Minimizing IV contrast exposure when appropriate
5. Treating severe anemia
6. Optimization of hemodynamics (Mean arterial BP>65mmHg).

The investigators plan to compare the results of this study with the historical data in the same patient population in the years of 7/1/2015-6/30/2017.

ELIGIBILITY:
Inclusion criteria:

* Adult patients that will undergo VAD placement.
* Patients able to give consent

Exclusion criteria:

* Patients on dialysis (hemodialysis or peritoneal dialysis)
* Non-elective VAD placement (VAD implantation decision made within 24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-02-17 (Actual); Study Completion 2019-02-17 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative AKI (within 5 post-op days) based on AKIN criteria | 5 days after the surgery
  The Acute Kidney Injury Network (AKIN) staging system has 3 stages: 1) serum creatinine increase ≥ 26.5 umol/L or increase to 1.5-2.0 fold from baseline, OR urine output <0.5 ml/kg/h for 6 h; 2) serum creatinine increase > 2.0-3.0 fold from baseline OR urine output <0.5 ml/kg/h for 12 h; 3) serum creatinine increase >3.0 fold from baseline OR serum creatinine ≥354 umol/l with an acute increase of at least 44 umol/l or need for Renal Replacement Therapy (RRT) OR urine output <0.3 ml/kg/h for 24 h OR anuria for 12 OR need for RRT

SECONDARY OUTCOMES:
Severity of postoperative AKI (within 5 post-op days) based on AKIN criteria | 5 days after the surgery
  The AKIN staging system has 3 stages: 1) serum creatinine increase ≥ 26.5 umol/L or increase to 1.5-2.0 fold from baseline, OR urine output <0.5 ml/kg/h for 6 h; 2) serum creatinine increase > 2.0-3.0 fold from baseline OR urine output <0.5 ml/kg/h for 12 h; 3) serum creatinine increase >3.0 fold from baseline OR serum creatinine ≥354 umol/l with an acute increase of at least 44 umol/l or need for Renal Replacement Therapy (RRT) OR urine output <0.3 ml/kg/h for 24 h OR anuria for 12 OR need for RRT
Length of hospital stay | 1 year after the surgery
  The length of hospital stay will be determined from the electronic medical record.
In hospital (perioperative) mortality and one-year mortality | Approximately 5 days after surgery, one year after enrollment
  The number of subjects who died in hospital (perioperatively) and one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qi Qian, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials